CLINICAL TRIAL: NCT05282979
Title: A Prospective, Single-arm Clinical Study Evaluating the Safety and Effectiveness of the Tixel Fractional System in the Treatment of Periorbital Wrinkles
Brief Title: A Prospective, Single Center, Single-Arm Clinical Study of 20 Participants to Reduce the Appearance of the Peri-orbital Wrinkles. Participants Will Receive up to Four Treatments With Tixel Every 4 Weeks. Follow-up Will Occur 1 Month and 3 Months Following Last Treatment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Physicians Laser and Dermatology Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLDI101
Record Dates: First submitted 2022-02-15; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Wrinkle
Keywords: Periorbital

STUDY DESIGN:
Intervention Model Description: All participates will undergo treatment with the Tixel 2 Device up to 4 treatments, 4 weeks apart and 2 Follow Up Visits
Masking Description: Blinded assessed of the improvement would be done between Last FU images and baseline, following randomization of the images.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tixel 2 (Experimental): Tixel 2 Treatment, 4 treatment sessions, followed by 2 Follow up sessions, 1 and 3 months after last treatment visit. Subject would be questioned about pain level, subjective downtime assessment and subjective response assessment. Images would be taken at the baseline and in Follow up visits.
  Interventions: Device: Tixel 2

INTERVENTIONS:
Device: Tixel 2 — Thermo-mechanical technology for fractional treatment of human skin. Dermal heating and coagulative effect that occur during the treatment session provide dermal remodeling and collagen restructuring that promote wrinkles appearance improvement.

SUMMARY:
A Prospective, Single center, Single-Arm Clinical Study of 13-20 study participants who are seeking a procedure to reduce the appearance of the peri-orbital wrinkles. Each study participant will receive up to four (4) treatments with the Tixel in a monthly interval. Follow-up will occur 1 month and 3 months following last treatment.

DETAILED DESCRIPTION:
A Prospective, Single center, Single-Arm Clinical Study of 13-20 participants who are seeking a procedure to reduce the appearance of the peri-orbital wrinkles, and meet study eligibility criteria, and have provided informed consent will be enrolled in the study. Each study participate will receive up to 4 treatments with Tixel in monthly interval. Follow-up will occur at 1 month and 3 months following the last visit.

The clinic visits will be as follow:

1. Base line (1st tx)
2. Phone-call visit (3 days after the first treatment)
3. 4 week (2nd tx)
4. 8 week (3rd tx)
5. 12 week (4th tx)
6. 4 weeks after the last treatment (1st Follow-up)
7. 12 weeks after the last treatment (2nd follow-up = 3 months follow-up, primary endpoint and the study completion visit)

Primary Safety Endpoint is the evaluation of related adverse events up to the 3-month visit after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 35-75 years old diagnosed with clinically evident fine (mild) to moderate depth periorbital wrinkles.
2. Willingness and ability to comply with all required study activities including returning for follow-up visits and protocol requirements.
3. The subject is able to provide written informed consent and perform the study's activities according to HIPAA guidelines.
4. Fitzpatrick wrinkle score of 3-7 in the peri-orbital areas per the treating investigator.
5. Stable body weight during the study period.
6. Skin Type I - V as per Fitzpatrick Skin Scale

Exclusion Criteria:

1. Past treatment with Tixel device.
2. The subject may not undergo treatment by the Tixel device according to the device's contra-indications for use, as defined in the User Manual and in the Instructions for Use and by any other labeling of the device.
3. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
4. Female subjects who are pregnant, or planning to become pregnant, or have given birth less than 3 months ago or are lactating.
5. Subjects with significant exposure to critical amounts of ultraviolet light (Suntan).
6. Subjects who have had the following treatments:

   1. a cosmetic procedure to improve periorbital rhytides within 6 months.
   2. Injectable filler in temples and in the upper face area to be treated within 12 months of investigation.
7. Any subject who have visible scars or other visible changes over the treated areas that may affect evaluation of response and/or quality of photography.
8. Subjects with any type of active cut, wound, inflammation, lesion (benign, premalignant or malignant) or active bacterial, viral, fungal, or herpetic infection on the skin on the designated treatment sites or in close proximity to it.
9. Existing or history of the following (when discussing skin conditions, refers only to the periorbital sites):

   1. skin malignancy, or any diagnosis of suspected malignancy
   2. Collagen or vascular or bleeding disease
   3. Immunosuppression or autoimmune disease
   4. History of persistent beyond 2 years post inflammatory hyperpigmentation.
   5. Active Acne Vulgaris, HSV-1, or any existing skin condition/disease that in the investigator's opinion would interfere with the evaluation of the safety of the study treatment and evaluation.
   6. Any skin condition which can induce bullous lesions, urticaria, or demonstrate a Koebner phenomenon (psoriasis, lichen planus, etc.).
   7. Any disease that inhibits pain sensation
   8. History of keloid formation.
   9. Conditions affecting healing rate (i.e. diabetes mellitus I or II, vascular condition, etc.)
   10. neuromuscular disorders
10. Subjects who have used, within 30 days, any medication over the periorbital area that can cause dermal hypersensitivity or affect skin characteristics over the treated area (i.e. topically applied retinoids, hydroquinone, Chemical peel of any strength: glycolic acid, lactic acid, salicylic acid)
11. Subjects who have used, systemic treatment which may induce dyspigmentation within 12 months, such as amiodarone, clofazinmine, minocycline or chloroquine.
12. Subjects currently taking or have taken an oral retinoid in the past 6 months;Subjects currently taking long-term oral steroid treatment.
13. Concurrent therapy that, in the principal investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study treatment.
14. Subjects who anticipate the need for major surgery or overnight hospitalization during the study that can affect the study schedule or treatment evaluation.
15. Enrollment in any active study involving the use of investigational devices or drugs which would impact the periorbital response.
16. Any other cause per the principal investigator's discretion.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
Safety Adverse Events report | Up to 12 months
  Evaluation of related adverse events up to the 3-month after last treatment visit
Effectiveness using Fitzpatrick Wrinkle Classification Scale (FWCS) | Up to 12 months
  Comparison of the proportion of subjects with a ≥ 1-score improvement on the Fitzpatrick Wrinkle Classification Scale (FWCS) at the 3-month visit compared to baseline. The FWCS is a clinically validated assessment tool used to assess skin wrinkle severity and elastosis on a scale from 1 through 9, where the lower score is considered better.

SECONDARY OUTCOMES:
Effectiveness using Fitzpatrick Wrinkle Classification Scale (FWCS)- Unblinded | Up to 12 months
  Assessment of improvement using Fitzpatrick Wrinkle Classification Scale (FWCS) at each visit compared to baseline by the handling physician. The FWCS is a clinically validated assessment tool used to assess skin wrinkle severity and elastosis on a scale from 1 through 9, where the lower score is considered better.
Effectiveness using GAIS-Global Aesthetic Improvement Scale Assessment-Unblinded | Up to 12 months
  Assessment of improvement using Global Aesthetic Improvement Scale Assessment at 1 month and 3 month follow up compared to baseline by the handling physician. Rating:
  1) Exceptional improvement patient; 2) Very improved patient; 3) Improved patient; 4)Unaltered patient; 5) Worsened patient
Evaluation of the pain and discomfort | Up to 12 months
  Evaluation of the pain and discomfort of the treatment as reported by the subject on a visual analog scale (VAS). Scoring will consist of making a mark on a 10-point scale. Each line will be awarded a score of 0-10 according to the level of pain when 0 is no pain and 10 is maximum pain possible.
Subject Subjective Downtime Assessment | Up to 12 months
  Evaluation of the period of time following the procedure during which the subject felt unable/unwilling to go out in public.
Patients' Reported Outcomes | Up to 12 months
  Subject Satisfaction Questionnaire and GAIS- Global Aesthetic Improvement Scale Assessment. Rating: 1) Exceptional improvement patient; 2) Very improved patient; 3) Improved patient; 4) Unaltered patient; 5) Worsened patient

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Garden, M.D., Principal Investigator — Physician Laser & Dermatology Institute
Locations (1):
- Physicians Laser & Dermatology Institute, LLC, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Background] Park SE, Kim SS, Kim CW, Her Y. A Prospective Split-Face Comparative Study of Periorbital Wrinkle Treatments: Fractional Erbium-Doped Yttrium Aluminum Garnet Laser, Intense Pulsed Light, and Topical 0.1% Tretinoin Cream. Ann Dermatol. 2016 Oct;28(5):650-652. doi: 10.5021/ad.2016.28.5.650. Epub 2016 Sep 30. No abstract available. PMID 27746652
- [Background] Manriquez JJ, Majerson Gringberg D, Nicklas Diaz C. Wrinkles. BMJ Clin Evid. 2008 Dec 16;2008:1711. PMID 19445782
- [Background] Gupta MA, Gupta AK. Photodamaged skin and quality of life; reasons for therapy. J Dermatol Treat 1996; 7:261-264
- [Background] Ganceviciene R, Liakou AI, Theodoridis A, Makrantonaki E, Zouboulis CC. Skin anti-aging strategies. Dermatoendocrinol. 2012 Jul 1;4(3):308-19. doi: 10.4161/derm.22804. PMID 23467476
- [Background] Hruza G, Taub AF, Collier SL, Mulholland SR. Skin rejuvenation and wrinkle reduction using a fractional radiofrequency system. J Drugs Dermatol. 2009 Mar;8(3):259-65. PMID 19271373
- [Background] Mulholland RS, Ahn DH, Kreindel M, Paul M. Fractional Ablative Radio-Frequency Resurfacing in Asian and Caucasian Skin: A Novel Method for Deep Radiofrequency Fractional Skin Rejuvenation. Journal of Cosmetics, Dermatological Sciences and Applications. 2012;2(3):144-150
- [Background] Michaud T, Gassia V, Belhaouari L. Facial dynamics and emotional expressions in facial aging treatments. J Cosmet Dermatol. 2015 Mar;14(1):9-21. doi: 10.1111/jocd.12128. Epub 2015 Jan 24. PMID 25620090
- [Background] Fitzpatrick RE, Goldman MP, Satur NM, Tope WD. Pulsed carbon dioxide laser resurfacing of photo-aged facial skin. Arch Dermatol. 1996 Apr;132(4):395-402. PMID 8629842
- [Background] Gold AH, Pozner J, Weiss R. A Fractional Bipolar Radiofrequency Device Combined with a Bipolar Radiofrequency and Infrared Light Treatment for Improvement in Facial Wrinkles and Overall Skin Tone and Texture. Aesthet Surg J. 2016 Oct;36(9):1058-67. doi: 10.1093/asj/sjw086. Epub 2016 Jul 29. PMID 27474769
- [Background] Kim JK, Roh MR, Park GH, Kim YJ, Jeon IK, Chang SE. Fractionated microneedle radiofrequency for the treatment of periorbital wrinkles. J Dermatol. 2013 Mar;40(3):172-6. doi: 10.1111/1346-8138.12046. Epub 2012 Dec 17. PMID 23252484
- See also: Causes of wrinkles and wrinkle prevention — http://www.mayoclinic.org/diseases-conditions/wrinkles/symptoms-causes/syc-20354927